CLINICAL TRIAL: NCT06664996
Title: Sintilimab Combined with Stereotactic Body Radiation Therapy As Neoadjuvant Therapy for Resectable Hepatocellular Carcinoma with Branch Portal Vein Tumor Thrombus: a Single-arm, Prospective Clinical Study
Brief Title: Sintilimab Combined SBRT As Neoadjuvant Therapy for Resectable HCC with PVTT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Wentao Wang, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-667
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Branch Portal Vein Tumor Thrombus
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment (Experimental): After obtaining informed consent, patients will undergo neoadjuvant therapy combining SBRT with sintilimab. SBRT will be administered on days 1, 3, and 5 at a dose of 8 Gy per fraction, totaling 3 fractions. Concurrently, patients will receive a first dose of sintilimab at 200 mg on day 1, followed by a second dose of 200 mg on day 22 (week 4, ±3 days). A radical hepatectomy is scheduled for day 50 (week 8, ±7 days). Tumor response will initially be evaluated using RECIST v1.1 criteria starting from the first administration, with a second pre-operative tumor imaging assessment at week 8 (±7 days). Post-surgery, patients will begin adjuvant treatment with sintilimab 200 mg every 3 weeks, continuing for 24 weeks. Follow-up assessments will occur every 3 months (±7 days) to collect data on disease status and survival, with a total follow-up duration of 1 year for each patient. This structured approach ensures precise timing and dosing while maintaining academic rigor and a logical sequen
  Interventions: Radiation: stereotactic body radiation therapy (SBRT); Drug: Sintilimab (approved)

INTERVENTIONS:
Radiation: stereotactic body radiation therapy (SBRT) — SBRT will be administered on days 1, 3, and 5 at a dose of 8 Gy per fraction, totaling 3 fractions.
Drug: Sintilimab (approved) — patients will receive a first dose of sintilimab at 200 mg on day 1, followed by a second dose of 200 mg on day 22 (week 4, ±3 days).

SUMMARY:
The goal of this single-arm, prospective clinical trial is to evaluate the safety and efficacy of neoadjuvant therapy combining sintilimab with stereotactic body radiation therapy (SBRT) in patients with resectable hepatocellular carcinoma (HCC) with branch portal vein tumor thrombus. The main questions it aims to answer are:

1. Is the combination of sintilimab and SBRT safe as neoadjuvant therapy?
2. How effective is this combination in treating resectable HCC with branch PVTT? Participants will be given a combination treatment of sintilimab and SBRT. Researchers will monitor their health conditions to assess the safety and effectiveness of this treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years, regardless of gender.
* Voluntary participation, as evidenced by signed informed consent, with the willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Diagnosis of hepatocellular carcinoma confirmed either histologically, cytologically, or based on characteristic imaging features (ultrasound, CT, MRI) and laboratory tests.
* Presence of measurable disease lesions per modified RECIST (mRECIST) criteria.
* Visible branch portal vein tumor thrombus (Japanese classification Vp1-Vp3 or Cheng's classification I-II) on imaging, deemed resectable after multidisciplinary consultation.
* No history of other malignancies.
* No prior treatments including targeted therapy, systemic chemotherapy, interventional treatments, surgical interventions, or radiotherapy before enrollment.
* Expected survival of at least 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Liver function classified as Child-Pugh A (score ≤6).
* Adequate organ and bone marrow function indicated by: serum creatinine ≤1.5 times the upper limit of normal, estimated glomerular filtration rate ≥50 mL/min/1.73m^2; total bilirubin ≤2 times the upper limit of normal; AST and ALT ≤2.5 times the upper limit of normal; AST/ALT ratio ≤3 times the upper limit of normal; platelet count ≥70×10^9/L, white blood cells count ≥3000/mm^3, and absolute neutrophil count ≥1500/mm^3 without transfusion to meet entry criteria.
* Female participants of childbearing potential must have a negative serum pregnancy test within 3 days prior to the commencement of the study medication, agree to use a highly effective method of contraception (e.g., intrauterine device, contraceptives, or condoms) during the study period and for 3 months after the last dose of study medication. Male participants with partners of childbearing potential must be surgically sterile or agree to use effective contraception during the study period and for 3 months after the last dose of study medication.

Exclusion Criteria:

* Previous treatments including interventional, immunotherapy, chemotherapy, or targeted therapy.
* Presence of confirmed distant metastasis on imaging or portal vein tumor thrombus involving the main portal vein (Vp4).
* Presence of refractory ascites or hepatic encephalopathy.
* Concurrent malignancy in other organs.
* Impaired organ function (hematologic, hepatic, renal) that precludes tolerance of treatment.
* Significant cardiac arrhythmias, myocardial ischemia, severe atrioventricular block, heart failure, or severe valvular heart disease.
* Severe bone marrow failure.
* Diagnosis of active autoimmune disease requiring any form of systemic treatment.
* Participation in another oncology clinical trial within the last 3 months.
* History of active tuberculosis or persistent, uncontrollable infections.
* Pregnant or breastfeeding participants.
* History of infection with the Human Immunodeficiency Virus (HIV).
* Any condition that, in the opinion of the investigator, would make participation in the study inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
1-year Disease-Free Survival (DFS) rate | DFS rate will be measured for each patient starting from the date they begin the treatment until one year after that date.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided